CLINICAL TRIAL: NCT01135940
Title: The Use of Dermabond vs. Standard Staple for Wound Closure in Children With Neuromuscular Scoliosis Undergoing Spinal Deformity Correction Surgery: A Phase II Study
Brief Title: The Use of Dermabond Versus Standard Staple for Wound Closure in Children With Neuromuscular Scoliosis Undergoing Spinal Deformity Correction Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: BCCH Telethon Grant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-00179
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Wounds
Keywords: neuromuscular scoliosis; dermabond; infection; wound closure
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 2-octylcyanoacrylate (Dermabond) closure
  Interventions: Device: 2-octylcyanoacrylate (Dermabond) closure
- 2 (Active Comparator): Standard staple closure
  Interventions: Device: Standard staple closure

INTERVENTIONS:
Device: 2-octylcyanoacrylate (Dermabond) closure — Standard procedure for closure of adipose/ subcutaneous layers. The subcuticular layer will be closed with a continuous 2-0 vicryl suture which will then be followed by Dermabond closure.
  Arms: 1
Device: Standard staple closure — Standard procedure for closure of adipose/ subcutaneous layers followed by staple closure
  Arms: 2

SUMMARY:
This is a prospective, Phase II (hypothesis generating) randomized pilot study investigating the efficacy of using Dermabond as a method of final wound closure as compared to the standard staple method in children with Neuromuscular Scoliosis undergoing spinal deformity correction surgery.

DETAILED DESCRIPTION:
1. To explore whether there is a difference in the incidence of wound infection in the Dermabond group vs. the skin staple group as measured by microbiological culture four days post-operatively. Wound infection is defined as prolonged sterile discharge (>4 days), positive wound cultures, or cellulitis four or more days post-operatively.
2. To explore whether there is a difference in the cosmetic result of the wound closure as measured by the Hollander wound evaluation scale. Our hypothesis is that the Dermabond group will have a better cosmetic result. Secondary outcome
3. To explore whether there is a difference in the time for final wound closure. Our hypothesis is that the Dermabond group will have a shorter time for final wound closure. Secondary outcome
4. To explore whether there is a difference in mean caregiver/parental satisfaction scores as measured by a visual analog scale. Our hypothesis is that parental satisfaction will be higher in the Dermabond group. Secondary outcome

ELIGIBILITY:
Inclusion Criteria:

* male or female 19 years or younger
* neuromuscular scoliosis
* undergoing posterior spinal instrumentation and fusion (one stage)

Exclusion Criteria:

* other non-neuromuscular causes of scoliosis
* previous history of spinal surgery
* previous incision over the operative site
* history of keloid formation
* allergy to superglue
* use of anticoagulation therapy

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Difference in the incidence of wound infection in Dermabond group versus the skin staple group | 12 weeks after surgery
  To explore whether there is a difference in the incidence of wound infection in Dermabond group versus the skin staple group as measured by microbiological culture taken 4 days post-operatively. Wound infection is defined as prolonged sterile discharge , positive wound cultures, or cellulitis four or more days post-operatively.

SECONDARY OUTCOMES:
Difference in the cosmetic result of the wound closure as measured by the Hollander wound evaluation scale | 12 weeks after surgery
  To explore whether there is a difference in the cosmetic result of the wound closure as measured by the Hollander wound evaluation scale. Our hypothesis is that the Dermabond group will have a better cosmetic result.
Difference in the time for final wound closure | Day of surgery
  To explore whether there is a difference in the time for final wound closure. Our hypothesis is that the Dermabond group will have a shorter time for final wound closure.
Difference in mean caregiver/parental satisfaction scores as measured by a visual analog scale | 12 weeks after surgery
  To explore whether there is a difference in mean caregiver/parental satisfaction scores as measured by a visual analog scale. Our hypothesis is that parental satisfaction will be higher in the Dermabond group.

CONTACTS AND LOCATIONS:
Overall Officials: Firoz Miyanji, MD, FRCSC, Principal Investigator — University of British Columbia; Christopher W. Reilly, MD, FRCSC, Study Director — University of British Columbia; Kishore Mulpuri, MBBS, MS, Study Director — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Department of Orthopaedics, Vancouver, British Columbia, Canada